CLINICAL TRIAL: NCT00307762
Title: Body-weight Supported Therapy Using Gait Trainer Versus Traditional Gait-oriented Physiotherapy in Acute Phase of Stroke. The Effectiveness of Gait Training and Brain Networks Using NBS (Navigating Brain Stimulation)
Brief Title: Gait Trainer vs Traditional Physiotherapy in Acute Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH5772732
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2008-01

CONDITIONS: Patients With Acute Stroke
Keywords: Stroke; Physiotherapy; Effectiveness; Gait trainer
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Gait trainer exercise actively for 20 minutes + 55 minutes other gait-oriented physiotherapy
  Interventions: Behavioral: intensified gait trainer
- 2 (Active Comparator): Overground walking exercises actively for 20 minutes + 55 minutes other gait-oriented physiotherapy
  Interventions: Behavioral: intensified gait trainer
- 3 (No Intervention): Control patients with ordinary therapy

INTERVENTIONS:
Behavioral: intensified gait trainer — Intensity and type of rehabilitation after stroke. Gait trainér + or overground walking + other gait-oriented physioteharpy. The third group (control patients) received traditional (ordinary) physiotherapy witn o efforts to intensify it.
  Arms: 1; 2

SUMMARY:
This is a trial aiming to evaluate the difference of effectiveness between two therapy methods in patients with acute stroke. The other aim is to use Navigated Brain Stimulation (NBS)to analyze changes in brain networks during the recovery and as the consequence of rehabilitation. The groups are:

* body-weight supported gate trainer rehabilitation
* gait-oriented traditional physiotherapy Patients in physiotherapy group will have 75 min physiotherapy daily every workday. This includes 20 minutes walking exercises in the traditional group while 20 minutes of gait trainer therapy in the gait trainer group. The evaluation of effectiveness of therapy in each group is made after three weeks' therapy and at six months. The goal is to have 40 patients until the end of June 2006.

DETAILED DESCRIPTION:
This study has been started in 2003 as a randomized study comparing rehabilitation with gait trainer and traditional gait-oriented physiotherapy.

* From the beginning of 2005, all patients have been evaluated using NBS (Navigating Brain Stimulation), a magnetic stimulation device. This stimulation is performed on day 3, 10 and 15 and at 6 months.

* The total number of patients recruited in the study is 57, seventeen (17) patients in gait trainer group and twenty (20) patients in the group of traditional physiotherapy. From the year 2005 onwards, ten (10 control patients have been recruited. Those patients have been selected with the exactly the same criteria as those who have been included in the treatment groups. The control patients have exactly the same evaluations at same time points, but their rehabilitation takes place according to the principles obeyed in the neurology clinic. Thus, they have not been randomised in any of the two treatment groups.
* Since the start of study, ten (10) patients have withdrawn from the study from various reasons (drop outs). One patient before randomization, 5 patients in the gait trainer group, one patient in the traditional physiotherapy group and 3 patients in the control group.
* Thus, the final group consists of 17 patients in the gait trainer group, 20 patients in the traditional therapy group and 10 patients in the control group.
* There will be 25 patients who have underwent the whole procedure of NBS: 9 patients in the gait trainer group, 8 patients in the traditional therapy group and 8 patients in the control group. The last 6-month follow-ups will take place in late August/early September 2007.

The idea of combining navigated magnetic brain stimulation (NBS)in the rehabilitation intervention study is to evaluate the change in brain networks during the recovery process, to see possible differences in these networks due to different rehabilitation methods and/or good vs. poor recovery. In connection with the magnetic stimulation, a 60-channel EEG map will be taken in order to measure the electrical spread of the induced neural electrical activity, which describes the state of the connections of the damaged brain area to other parts of the brain as well as of possible activation of new neural connections.

This arrangement allows a unique opportunity to study the re-organisation of brain structures after stroke and brain plasticity in general in recovering brain.

For the evaluation of functional recovery, a combination of relevant scales of motor function will be measured during the study. Those are: Rivermead Mobility Index, Rivermead Motor Assessment , Modified Motor Assessment Scale, Functional ambulation Category, Physical Cost Index, 6-minute walking time. In addition, Barthel index, Scandinavian Stroke Scale and NIH Scale will be performed in the beginning and at the end.

ELIGIBILITY:
Inclusion Criteria:

* Supratentorial stroke within 8 days of onset
* Barthel index 25-75

Exclusion Criteria:

* Severe cognitive disorder
* Severe cardiac disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2003-05; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Improvement ín motor function among patients in each group

SECONDARY OUTCOMES:
Modified Motor Assessment Scale (MMAS)
Rivermead Motor Assessment Scale (RMA)
Rivermead Mobility Index (RMI)
Ten meters walking time (10MWT)
Six-min walking distance
Barthel index
NIHSS

CONTACTS AND LOCATIONS:
Overall Officials: Sivenius MR Sivenius, MD, PhD, Study Director — Department of Neurology, Kuopio University Hospital
Locations (1):
- Department of Neurology, University Hospital of Kuopio, Kuopio, Finland

REFERENCES:
- [Derived] Peurala SH, Airaksinen O, Jakala P, Tarkka IM, Sivenius J. Effects of intensive gait-oriented physiotherapy during early acute phase of stroke. J Rehabil Res Dev. 2007;44(5):637-48. doi: 10.1682/jrrd.2006.05.0039. PMID 17943675